CLINICAL TRIAL: NCT00414466
Title: A Randomized Double Blind, Placebo-controlled, Dose Response Study of Intraspinal Gabapentin (MDT2004) in Subjects With Chronic, Intractable Pain.
Brief Title: A Safety and Effectiveness Study of Intraspinal Gabapentin (MDT2004) for the Treatment of Chronic Pain
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study closed and subject follow-up completed following analysis of blinded study data.
Sponsor: MedtronicNeuro (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1622
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Results first posted 2011-06-08 (Estimated); Last update posted 2013-08-23 (Estimated); Status verified 2013-08

CONDITIONS: Chronic Intractable Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (0mg/day) (Placebo Comparator): Intraspinal Placebo delivered continuously for 29 days via an implantable infusion system
  Interventions: Drug: Intraspinal Gabapentin
- Gabapentin Low (1mg/day) (Active Comparator): Intraspinal Gabapentin Low delivered continuously for 22 days via an implantable infusion system followed by 7 days infusion at half dose
  Interventions: Drug: Intraspinal Gabapentin
- Gabapentin Medium (6mg/day) (Active Comparator): Intraspinal Gabapentin Medium delivered continuously for 22 days via an implantable infusion system followed by 7 days infusion at half dose
  Interventions: Drug: Intraspinal Gabapentin
- Gabapentin High (30mg/day) (Active Comparator): Intraspinal Gabapentin High delivered continuously for 22 days via an implantable infusion system followed by 7 days infusion at half dose
  Interventions: Drug: Intraspinal Gabapentin

INTERVENTIONS:
Drug: Intraspinal Gabapentin — Surgical implantation of a drug infusion system with intrathecal (spinal) delivery of active drug (1 of 3 possible dose levels) or placebo (saline) for 22 days followed by 7 days of infusion at half dose level. Subjects may then continue in open-label treatment with study drug. Dosage in open-label may be adjusted to meet subject needs.

SUMMARY:
The purpose of this study is to determine the safety and minimum effective dose of intraspinal gabapentin when delivered through an implanted drug infusion system.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain below the neck present for a minimum of one year.
* Diagnosis of at least one of the following:

  * back pain with or without leg pain,
  * post-herpetic neuralgia,
  * complex regional pain syndrome (CRPS) 1 or 2,
  * diabetic neuropathy,
  * or a general neuropathic condition; medically stable and able to undergo surgery for implantation of the drug infusion system.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Actual)
Dates: Start 2006-12; Primary Completion 2009-12 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Innovative Spine Care, Little Rock, Arkansas
  - Napa Pain Institute, Napa, California
  - Sarasota Pain Medicine Research, Sarasota, Florida
  - WK River Cities Clinical Research Center, Shreveport, Louisiana
  - MAPS Applied Research Center, Edina, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - U B Neurosurgery, Inc., Buffalo, New York
  - The Center for Clinical Research, Winston-Salem, North Carolina
  - Pain Research of Oregon, LLC, Eugene, Oregon
  - Oregon Health & Science University, Neurosurgery Department, Portland, Oregon
  - Lehigh Valley Hospital Center for Pain Management, Allentown, Pennsylvania
  - Pinnacle Pain Medicine, Dallas, Texas
  - Axis Spine Care/Texas Spine & Joint, Tyler, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah

REFERENCES:
- [Derived] Rauck R, Coffey RJ, Schultz DM, Wallace MS, Webster LR, McCarville SE, Grigsby EJ, Page LM. Intrathecal gabapentin to treat chronic intractable noncancer pain. Anesthesiology. 2013 Sep;119(3):675-86. doi: 10.1097/ALN.0b013e3182a10fbf. PMID 23835590

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 254 subjects were enrolled into the study between December 2006 and October 2009.
Pre-assignment Details: During a 2-week screening period subjects were required to meet eligibility criteria including maintaining stable pain medications and demonstrating a numerical pain rating score of 6 or greater averaged over the last 7 days of screening. A total of 170 subjects met eligibility criteria, were implanted with an infusion system and were randomized.
Groups:
- 1 Placebo (0mg/Day): Intraspinal Placebo delivered continuously for 29 days via an implantable infusion system
- 2 Gabapentin Low (1mg/Day): Intraspinal Gabapentin Low (1mg/day) delivered continuously for 22 days via an implantable infusion system followed by 7 days of infusion at half dose
- 3 Gabapentin Medium (6mg/Day): Intraspinal Gabapentin Medium (6mg/day) delivered continuously for 22 days via an implantable infusion system followed by 7 days of infusion at half dose
- 4 Gabapentin High (30mg/Day): Intraspinal Gabapentin High (30mg/day) delivered continuously for 22 days via an implantable infusion system followed by 7 days of infusion at half dose
Period: Overall Study
Arm/Group | 1 Placebo (0mg/Day) | 2 Gabapentin Low (1mg/Day) | 3 Gabapentin Medium (6mg/Day) | 4 Gabapentin High (30mg/Day)
Started | 44 | 42 | 41 | 43
Completed | 42 | 42 | 40 | 42
Not Completed | 2 | 0 | 1 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0
Not completed — Withdrawn by Sponsor | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 1 Placebo: Intraspinal Placebo delivered continuously for 29 days via an implantable infusion system
- 2 Gabapentin Low: Intraspinal Gabapentin Low delivered continuously for 22 days via an implantable infusion system followed by 7 days of infusion at half dose
- 3 Gabapentin Medium: Intraspinal Gabapentin Medium delivered continuously for 22 days via an implantable infusion system followed by 7 days of infusion at half dose
- 4 Gabapentin High: Intraspinal Gabapentin High delivered continuously for 22 days via an implantable infusion system followed by 7 days of infusion at half dose
- Total: Total of all reporting groups
Arm/Group | 1 Placebo | 2 Gabapentin Low | 3 Gabapentin Medium | 4 Gabapentin High | Total
Number analyzed (Participants) | 44 | 42 | 41 | 43 | 170
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 39 | 41 | 40 | 40 | 160
  >=65 years | 5 | 1 | 1 | 3 | 10
Age Continuous [Mean (Standard Deviation); unit: years] | 51.8 (11.2) | 50.1 (9.9) | 48.1 (9.4) | 48.3 (11.1) | 49.6 (10.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 28 | 20 | 23 | 98
  Male | 17 | 14 | 21 | 20 | 72
Region of Enrollment [Number; unit: participants]
  United States | 44 | 42 | 41 | 43 | 170

OUTCOME MEASURES:

1. Primary Outcome: Changes in a Pain Rating Scale After 3 Weeks of Blinded Treatment.
Description: Average pain score calculated over last 7 days of baseline minus average pain score calculated over last 7 days of follow-up using the Numeric Pain Rating Scale where 0=no pain, 10=worst possible pain.
Time Frame: Baseline and Post-randomization Day 22
Population: Primary efficacy analysis was performed on the 167 randomized subjects that completed at least 4 days of the electronic pain diary during the last 7 days prior to the Day 22 or Early Termination Visit as per protocol. No imputation methods were used.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- 2 Gabapentin Low: Intraspinal Gabapentin Low (1mg/day) delivered continuously for 22 days via an implantable infusion system followed by 7 days of infusion at half dose
- 3 Gabapentin Medium: Intraspinal Gabapentin Medium (6mg/day) delivered continuously for 22 days via an implantable infusion system followed by 7 days of infusion at half dose
- 4 Gabapentin High: Intraspinal Gabapentin High (30mg/day) delivered continuously for 22 days via an implantable infusion system followed by 7 days of infusion at half dose
Arm/Group | 1 Placebo | 2 Gabapentin Low | 3 Gabapentin Medium | 4 Gabapentin High
Number analyzed (Participants) | 43 | 42 | 41 | 41
Scores on a scale | 0.48 (1.52) | 0.40 (1.33) | 0.10 (0.99) | -0.02 (1.11)
Statistical Analysis 1: Comparison: 1 Placebo vs 2 Gabapentin Low; Williams' test for Minimum Effective Dose was used to compare each active group to the placebo; Test type: Superiority or Other; p = 0.802, Williams test for minimum effective dose — The a priori threshold for statistical significance was 0.05, two-sided
Statistical Analysis 2: Comparison: 1 Placebo vs 3 Gabapentin Medium; Williams' test for Minimum Effective Dose was used to compare each active group to the placebo; Test type: Superiority or Other; p = 0.874, Williams test for minimum effective dose — The a priori threshold for statistical significance was 0.05, two-sided
Statistical Analysis 3: Comparison: 1 Placebo vs 4 Gabapentin High; Williams' test for Minimum Effective Dose was used to compare each active group to the placebo; Test type: Superiority or Other; p = 0.899, Williams test for minimum effective dose — The a priori threshold for statistical significance was 0.05, two-sided

2. Secondary Outcome: Responder Analysis Between Active Treatment and Placebo Groups.
Description: Responders were subjects that reported at least a 30% decrease in average daily pain scores between baseline and Day 22.
Time Frame: Baseline to Post-randomization Day 22
Population: All 170 randomized subjects were included as per protocol. Subjects experiencing an intolerable adverse event, discontinuing due to an adverse event or lack of efficacy, or not providing data were considered non-responders.
Measure: Number; unit: Participants
Arm/Group | 1 Placebo | 2 Gabapentin Low | 3 Gabapentin Medium | 4 Gabapentin High
Number analyzed (Participants) | 44 | 42 | 41 | 43
Participants | 4 | 4 | 1 | 2
Statistical Analysis 1: Comparison: 1 Placebo vs 2 Gabapentin Low; Test type: Superiority or Other; p = 1.000, Fisher Exact — The a priori threshold for statistical significance was 0.05, two-sided. Hochberg's adjustment for multiple comparisons was used
Statistical Analysis 2: Comparison: 1 Placebo vs 3 Gabapentin Medium; Test type: Superiority or Other; p = 1.000, Fisher Exact — [p-value comment as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: 1 Placebo vs 4 Gabapentin High; Test type: Superiority or Other; p = 1.000, Fisher Exact — [p-value comment as in outcome 2, analysis 1]

3. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events
Description: Evaluation of adverse event profiles between placebo and active treatment groups.
Time Frame: Randomization to Post-randomization Day 29 (includes dose reduction)
Population: All randomized subjects were included as per protocol.
Measure: Number; unit: Participants
Arm/Group | 1 Placebo | 2 Gabapentin Low | 3 Gabapentin Medium | 4 Gabapentin High
Number analyzed (Participants) | 44 | 42 | 41 | 43
Participants | 40 | 32 | 37 | 36
Statistical Analysis 1: Comparison: 1 Placebo vs 2 Gabapentin Low; Test type: Superiority or Other; p = 0.083, Fisher Exact — The a priori threshold for statistical significance was 0.05, two-sided. No adjustments for multiple comparisons were used
Statistical Analysis 2: Comparison: 1 Placebo vs 3 Gabapentin Medium; Test type: Superiority or Other; p = 1.000, Fisher Exact — [p-value comment as in outcome 3, analysis 1]
Statistical Analysis 3: Comparison: 1 Placebo vs 4 Gabapentin High; Test type: Superiority or Other; p = 0.352, Fisher Exact — [p-value comment as in outcome 3, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse events are reported through 29 days post-randomization, including 22 days of dosing at the randomized dose and 7 days of dose reduction.
Description: All randomized subjects were included in adverse event summaries.
Arm/Group | 1 Placebo | 2 Gabapentin Low | 3 Gabapentin Medium | 4 Gabapentin High
Serious Adverse Events (participants affected / at risk) | 1/44 | 1/42 | 4/41 | 4/43
Other Adverse Events (participants affected / at risk) | 30/44 | 21/42 | 27/41 | 25/43
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Placebo (N=44) | 2 Gabapentin Low (N=42) | 3 Gabapentin Medium (N=41) | 4 Gabapentin High (N=43)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Implant site infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bone marrow disorder (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neuropathic pain (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oesophageal spasm (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Closed head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Therapeutic agent toxicity (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 1 Placebo (N=44) | 2 Gabapentin Low (N=42) | 3 Gabapentin Medium (N=41) | 4 Gabapentin High (N=43)
Implant site infection (Infections and infestations) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
Influenza (Infections and infestations) | 2 (2) | 1 (1) | 0 (0) | 4 (4)
Nasopharyngitis (Infections and infestations) | 3 (3) | 1 (1) | 2 (2) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 2 (2) | 1 (1) | 3 (3) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 3 (3)
Insomnia (Psychiatric disorders) | 2 (3) | 1 (1) | 3 (3) | 2 (2)
Dizziness (Nervous system disorders) | 1 (1) | 3 (3) | 6 (6) | 4 (4)
Headache (Nervous system disorders) | 6 (6) | 4 (4) | 5 (5) | 3 (3)
Somnolence (Nervous system disorders) | 4 (4) | 1 (1) | 2 (2) | 4 (4)
Nausea (Gastrointestinal disorders) | 4 (4) | 4 (4) | 4 (4) | 5 (5)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (7) | 5 (5) | 2 (2) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (3) | 4 (4) | 1 (1) | 3 (3)
Fatigue (General disorders) | 3 (3) | 1 (1) | 3 (3) | 3 (3)
Oedema Peripheral (General disorders) | 1 (1) | 0 (0) | 2 (2) | 4 (4)
Pain (General disorders) | 3 (3) | 4 (4) | 6 (7) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less